CLINICAL TRIAL: NCT01725919
Title: Examining Mechanisms of Neuroplasticity Following Motor Rehabilitation in Stroke
Brief Title: Examining How Motor Rehabilitation Promotes Brain Reorganization Following Stroke, an MRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Yousef Hannawi, Assistant Professor- Neurology, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 60034699
Record Dates: First submitted 2012-11-06; First posted 2012-11-14 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Hemiparesis
Keywords: motor; stroke; hemiparesis; rehabilitation; constraint induced movement therapy; CI therapy
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate CI therapy (Experimental)
  Interventions: Behavioral: CI therapy
- Delayed CI therapy (Active Comparator)
  Interventions: Behavioral: CI therapy

INTERVENTIONS:
Behavioral: CI therapy — constraint induced movement therapy

SUMMARY:
Constraint-induced movement therapy (CI therapy) is a highly efficacious treatment for residual motor disability in chronic stroke. Its effectiveness is believed to be due, at least in part, to the therapy's ability to aid the brain in "rewiring itself." For example, CI therapy produces increases in the amount of grey matter (the parts of the brain where neuron cell bodies are most closely clustered) in certain areas of the human brain (Gauthier et al., 2008). The cellular and molecular mechanisms that are responsible for this increase in grey matter volume are not known, however. Thus, it is unclear how the therapy helps brains "rewire" themselves. This study aims to better understand the timecourse and cellular/molecular nature of brain changes during CI therapy. Because there is currently no way to directly measure cellular/molecular changes in the brain noninvasively, this study will infer what is happening on a microstructural level using new MRI techniques (three dimensional pictures of the brain). For example, by charting the timecourse of grey matter changes during CI therapy, and cross-comparing this to what is known about the timecourses of different cellular/molecular processes, the investigators can gain a greater understanding of what cellular processes may be responsible for increases in grey matter. The investigators will gain additional information about which cellular processes are important for rehabilitation-induced improvement by measuring larger-scale changes (e.g., amount of blood flow through different brain areas) that accompany cellular changes. The investigators are hopeful that by better understanding how CI therapy can change the brain, the effectiveness of rehabilitation can be improved upon. For example, insight into the mechanisms of rehabilitation-induced brain change may suggest particular drug targets to increase brain plasticity. This study will help us better understand how the brain repairs itself after injury.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age and over
* Experienced a stroke resulting in mild to moderate hemiparesis (some residual motor function, e.g. able to pick up a washcloth placed flat on a table) at least 6 months prior to enrollment. Suggested active range of motion criteria for this level of impairment include: 45° shoulder abduction and flexion, 20° elbow extension, 20° wrist extension, and 10° extension of thumb and fingers.
* Preserved ability to comprehend and participate in basic elements of the therapy

Exclusion Criteria:

* Concurrent participation in other experimental trials for treatment of motor dysfunction
* Having received botulinum toxin injection within the past 3 months
* Previous intensive rehabilitation in the chronic phase post-stroke
* Serious/uncontrolled medical problems (e.g., dementia, severe pain, end-stage or degenerative diseases)
* Kidney disease as evidenced by eGFR<60
* Anemia
* Sickle cell disease
* History of kidney transplant
* Other evidence/history of renal disease
* Pregnancy
* Implanted metallic parts of implanted electronic devices, including pacemakers, defibrillators, aneurism clip or implant medication pump that are MRI incompatible
* An implanted brain stimulator
* Permanent tattoo (e.g., eye liner) containing metallic coloring
* Claustrophobia precluding MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Brain structure | Participants will be followed for 4-6 weeks. Change in brain structure at mid-treatment (after 1 week of CI therapy), post-treatment (after 2 weeks of therapy), and at 2-week follow-up will be measured.
  Assessed via dynamic susceptibility contrast MRI, diffusion tensor MRI, MRI-based myelin mapping, T1-weighted MRI

SECONDARY OUTCOMES:
Motor function | Participants will be followed for 4-6 weeks. Change in motor function at mid-treatment (after 1 week of CI therapy), post-treatment (after 2 weeks of therapy), and at 2-week follow-up will be measured.
  Assessed via Wolf Motor Function Test, Action Research Arm Test, Motor Activity Log

CONTACTS AND LOCATIONS:
Overall Officials: Yousef Hannawi, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Rafiei MH, Kelly KM, Borstad AL, Adeli H, Gauthier LV. Predicting Improved Daily Use of the More Affected Arm Poststroke Following Constraint-Induced Movement Therapy. Phys Ther. 2019 Dec 16;99(12):1667-1678. doi: 10.1093/ptj/pzz121. PMID 31504952
- [Derived] Kelly KM, Borstad AL, Kline D, Gauthier LV. Improved quality of life following constraint-induced movement therapy is associated with gains in arm use, but not motor improvement. Top Stroke Rehabil. 2018 Oct;25(7):467-474. doi: 10.1080/10749357.2018.1481605. Epub 2018 Sep 22. PMID 30246613